CLINICAL TRIAL: NCT01341210
Title: The Study of the Knowledge, Attitudes, and Decision Making Towards Clinical Trials in Cancer Patients
Brief Title: Observational Study of the Decision Making Towards Clinical Trials in Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, National Taiwan University Hospital, National Taiwan University Hospital
Other Study IDs: 201101071RC
Record Dates: First submitted 2011-04-21; First posted 2011-04-25 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Lung Cancer; Liver Cancer
Keywords: Patients Satisfaction; Decision Making; Informed Consent
MeSH Terms: conditions — Lung Neoplasms; Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a cross-sectional, observational and correlational survey study.This study is aim to survey the the knowledge, attitudes, and decision making towards clinical trials in cancer patients in Taiwan (R.O.C.), which attempts to invite some cancer patients who have been experienced the treatment clinical trials' informed consent process. The research tool is a questionnaire which includes some scale: (1)Clinical trial Knowledge scale, (2) Attitude toward randomized clinical trials scale, (3) Shared Decision Making(SDM-Q-9),(4) Satisfaction with Decision (SWD-scale), and (5) Decision Regret scale(DRS). The investigators expect the research outcome can provide some instructions to improve patients' autonomy, satisfaction of the decision making and communication process between patients and Medical professors whenever cancer patients participating in clinical trials.

DETAILED DESCRIPTION:
This study is been conduct in National Taiwan University Hospital , Taiwan. The main measurement tool is a self-report questionnaire, which is designed to answer some outcome measures for the following aspect:

1. To find out the knowledge, attitudes, shared decision making level, subjective norm, and behavior intentions towards clinical trials in cancer patients.
2. To find out the main influencing factors of behavior intentions towards participating in clinical trials

ELIGIBILITY:
Inclusion Criteria:

1. Cancer patients who have been approved lung cancer or liver cancer.
2. Patients who have been experienced the Informed consent process about clinical trial, which duration is in 6 months before they enter this study.

Exclusion Criteria:

1. Patients who have conscious disorientation that can not answer questionnaire
2. Patients only participate in some Gene clinical trials without treatment or drugs.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, cancer patients who have experience in contact with clinical trials
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2011-02; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
The influencing factors of behavior intentions towards participating in clinical trials | in 24 months
  The influencing factors was defined as following measurement scale:
  1. Knowledge
  2. Attitude
  3. decision making process
  4. sex
  5. age
  6. education

SECONDARY OUTCOMES:
The knowledge towards clinical trials in cancer patients | 24 months
The attitudes towards clinical trials in cancer patients | in 24 months
The shared decision making level towards clinical trials in cancer patients | 24 months
The subjective norm and behavior intentions towards clinical trials in cancer patients | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Yu Hu, PHD, Principal Investigator — National Taiwan University, Department of Nursing
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan